CLINICAL TRIAL: NCT04214249
Title: BLockade of PD-1 Added to Standard Therapy to Target Measurable Residual Disease in Acute Myeloid Leukemia 1 (BLAST MRD AML-1): A Randomized Phase 2 Study of the Anti-PD-1 Antibody Pembrolizumab in Combination With Conventional Intensive Chemotherapy as Frontline Therapy in Patients With Acute Myeloid Leukemia
Brief Title: BLAST MRD AML-1: BLockade of PD-1 Added to Standard Therapy to Target Measurable Residual Disease in Acute Myeloid Leukemia 1- A Randomized Phase 2 Study of Anti-PD-1 Pembrolizumab in Combination With Intensive Chemotherapy as Frontline Therapy in Patients With Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-08626; NCI-2019-08626 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2000028858; 10300 (Other: Yale University Cancer Center LAO); 10300 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Acute Myeloid Leukemia Post Cytotoxic Therapy; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; Cytarabine; Daunorubicin; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Idarubicin; 4-demethoxydaunorubicin bis(hydrazone); pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (cytarabine, idarubicin, daunorubicin, HSCT) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Hematopoietic Cell Transplantation; Drug: Idarubicin Hydrochloride; Procedure: Multigated Acquisition Scan; Biological: Pembrolizumab; Procedure: Punch Biopsy
- Arm II (cytarabine, idarubicin, daunorubicin, HSCT) (Active Comparator): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Hematopoietic Cell Transplantation; Drug: Idarubicin Hydrochloride; Procedure: Multigated Acquisition Scan; Procedure: Punch Biopsy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cytarabine — Given via continuous IV infusion
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Hematopoietic Cell Transplantation — Undergo HSCT
  Other Names: HCT; Hematopoietic Stem Cell Infusion; HEMATOPOIETIC STEM CELL TRANSPLANT; Hematopoietic Stem Cell Transplantation; HSCT; SCT; Stem Cell Transplant; stem cell transplantation; Stem Cell Transplantation, NOS
Drug: Idarubicin Hydrochloride — Given IV
  Other Names: Idamycin; Idamycin PFS; Idarubicin HCl; IMI-30; SC-33428; Zavedos
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Arm I (cytarabine, idarubicin, daunorubicin, HSCT)
Procedure: Punch Biopsy — Undergo a skin punch biopsy
  Other Names: BIOPSY, PUNCH; Punch Biopsy of Skin

SUMMARY:
This phase II trial studies how well cytarabine and idarubicin or daunorubicin with or without pembrolizumab work in treating patients with newly-diagnosed acute myeloid leukemia. Chemotherapy drugs, such as cytarabine, idarubicin, and daunorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving induction chemotherapy with pembrolizumab may work better than induction chemotherapy alone in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the percentage of patients with minimal residual disease (MRD) negative complete remission (CR) (MRD-CR), or with minimal residual disease (MRD) negative complete remission with incomplete recovery (CRi) (MRD-CRi) as measured by flow cytometry at the end of first cycle of consolidation therapy with chemotherapy + pembrolizumab (MK-3475) and compare between the two study arms.

SECONDARY OBJECTIVES:

I. Assess the rate of complete remission (CR)/complete remission with incomplete count recovery (CRi) as defined per European Leukemia Net 2017 response criteria at time of count recovery after induction therapy with chemotherapy + pembrolizumab (MK-3475) (Dohner et al., 2017).

II. Rates of complete remission with partial recovery count (CRh) and hematologic improvement (HI) to red blood cells and platelets.

III. Assess the rates of MRD negativity at day 14, MRD-negative CR at end of induction therapy and MRD negative CR after last consolidation cycle.

IV. Assess event free survival (EFS), measured from randomization to failure to achieve CR/CRi, relapse or death from any cause, and relapse free survival (RFS), calculated as the time from first documentation of CR/CRi to either disease relapse or death from any cause.

V. Assess the duration of response (DOR, defined as the time from first CR/CRi to the date of the first documented relapse or death, whichever occurs first) and overall survival (OS), defined as time from randomization to death from any cause.

VI. Assess safety endpoints including proportion of patients who develop severe toxicity as defined in the protocol.

EXPLORATORY OBJECTIVES:

I. MRD assessment by duplex sequencing (DS) and comparing DS and multiparameter flow cytometry for MRD detection as an exploratory biomarker.

II. Assessment of immune-checkpoint expression and dynamic change of immune cell subsets in response to the combination of checkpoint-inhibition and backbone combination in acute myeloid leukemia (AML).

III. High-throughput sequencing of the T-cell receptor (TCR) Vb CDR3 regions on ﬂow cytometrically sorted t-cell subsets to assess the effect of immunotherapy on the diversity of the t-cell repertoire and assess for correlation to clinical outcomes.

IV. Investigation of protein signatures and ribonucleic acid (RNA) signatures associated with response and efficacy using O-link cytokine panel and RNA-sequencing (seq), respectively.

V. Determination of mutational load by whole exome sequencing to assess for correlation with clinical outcomes, immune infiltrating profile, and T cell repertoire diversity and clonality.

VI. Correlate gut microbiome at baseline and changes in the microbiome with clinical response, both in standard chemotherapy and immunotherapy/chemotherapy therapy settings.

VII. MRD assessment using duplex sequencing strategy for circulating cell-free tumor deoxyribonucleic acid (DNA) and correlation with long-term outcomes.

OUTLINE: Patients are randomized to 1 of 2 arms.

INDUCTION PHASE:

ARM I: Patients receive cytarabine via continuous intravenous (IV) infusion on days 1-7 and idarubicin hydrochloride IV over 15-30 minutes or daunorubicin hydrochloride IV over 15-30 minutes on days 1-3 of a 28-35 day cycle. Patients who have evidence of residual leukemia receive cytarabine via continuous IV infusion over days 1-5 and idarubicin hydrochloride IV over 15-30 minutes or daunorubicin hydrochloride IV over 15-30 minutes on days 1-2 for an additional cycle in the absence of disease progression or unacceptable toxicity. Beginning day 8, patients receive pembrolizumab IV over 25-40 minutes. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve a CR or a CRi may undergo hematopoietic stem cell transplantation (HSCT) per physician discretion or continue to consolidation therapy.

ARM II: Patients receive cytarabine via continuous IV infusion on days 1-7 and idarubicin hydrochloride IV over 15-30 minutes or daunorubicin hydrochloride IV over 15-30 minutes on days 1-3 of a 28-35 day cycle. Patients who have evidence of residual leukemia receive cytarabine via continuous IV infusion over days 1-5 and idarubicin hydrochloride IV over 15-30 minutes or daunorubicin hydrochloride IV over 15-30 minutes on days 1-2 for an additional cycle in the absence of disease progression or unacceptable toxicity. Patients who achieve a CR or a CRi may undergo HSCT per physician discretion or continue to consolidation therapy.

CONSOLIDATION THERAPY:

ARM I: Within 4 weeks of remission status documentation, patients receive high-dose cytarabine (HiDAC) IV over 1-3 hours every 10-12 hours on days 1, 3, and 5 for a total of 6 doses and pembrolizumab IV over 25-40 minutes. Cycles with HiDAC repeat every 28-42 days and cycles with pembrolizumab repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who remain in CR or CRi receive up to 3 additional cycles of HiDAC and pembrolizumab in the absence of disease progression or unacceptable toxicity and continue to maintenance therapy.

ARM II: Within 4 weeks of remission status documentation, patients receive HiDAC IV over 1-3 hours every 12 hours on days 1, 3, and 5 for a total of 6 doses in the absence of disease progression or unacceptable toxicity. Patients who remain in CR or CRi receive up to 3 additional cycles of HiDAC in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY:

ARM I: Patients receive pembrolizumab IV over 25-40 minutes. Cycles repeat every 3 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

All patients also undergo a skin punch biopsy during screening and undergo bone marrow biopsy and aspiration, collection of blood samples, and echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening and on study. Patients may optionally undergo computed tomography (CT) scan during screening.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for up to 5 years. Patients who undergo HSCT are also followed up at 100 days post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and pathologically-confirmed AML, confirmed by a bone marrow aspirate and/or biopsy and/or peripheral blood with >= 20% myeloid blasts. Bone marrow biopsy, or aspirate or peripheral blood that were obtained up to 3 weeks before signing consent are allowed for purposes of confirming AML diagnosis for eligibility purposes. Secondary AML (that is arising from prior myelodysplastic syndrome [MDS] as well as therapy-related [t]-AML) are also allowed. Clarifications: AML arising from myeloproliferative neoplasms (MPN), MPN/MDS overlap (including chronic myelomonocytic leukemia [CMML]) or another myeloid malignancy are NOT allowed. Note 1: Patients must have evidence of bone marrow involvement on aspirate or biopsy. Patients with only extramedullary disease and no bone marrow involvement will be excluded. Note 2: Every effort should be made to get an aspirate for central flow assessment at screening and all subsequent required time points, but in cases where an aspirate cannot be collected-including dry taps-the patient will not be excluded and assessments will be performed on peripheral blood (PB) which should be collected at every time that bone marrow (BM) is collected. Note 3: Some patients with AML require initiation of therapy quickly after diagnosis, and full metaphase karyotype results in some centers can take 2-3 weeks to result. To avoid this issue being an impediment to accrual to study or to cause delays in initiation of therapy in patients who need fast initiation of therapy, we allow use of karyotype and/or fluorescence in situ hybridization (FISH) results (as well as FLT3 results) on samples from blood or marrow that were obtained up to 3 weeks before signing consent for purposes of eligibility and stratification. In any case, results from FISH or karyotype should show if core-binding factor (CBF) abnormalities are present by time of randomization as the presence of CBF abnormalities is a required stratification factor
* Age >= 18 and =< 75 years

  * Because no dosing or adverse event (AE) data are currently available on the use of pembrolizumab (MK-3475) in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< -2
* The patient has to be eligible to receive intensive "7+3" induction chemotherapy as judged by the treating physician
* Prior use of hypomethylating agents (HMA), lenalidomide, erythropoiesis-stimulating agents (ESAs), and growth factors is allowed if used to treat prior MDS. AML must be previously untreated except as outlined below (hydroxyurea, or tretinoin [ATRA], or leukapheresis). Note: One dose of prophylactic intrathecal therapy is allowed during or before screening if a lumbar puncture is performed to rule out central nervous system (CNS) involvement
* Hydroxyurea/leukapheresis allowed for control of hyperleukocytosis but hydroxyurea must be discontinued day prior to start of chemotherapy
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (CrCl) >= 60 mL/min for patient with creatinine levels > 1.5 x institutional ULN (within 3 days prior to the first day of 7+3)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
  * Glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl
* Total bilirubin =< 1.5 x ULN or direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 x ULN (within 3 days prior to the first day of 7+3)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN OR =< 5 x ULN for patients with liver metastases (within 3 days prior to the first day of 7+3)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 3 days prior to the first day of 7+3)
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (within 3 days prior to the first day of 7+3)
* Patients with a known history of being human immunodeficiency virus (HIV) positive may participate IF they meet the following eligibility requirements:

  * They must be stable on their anti-retroviral regimen, and they must be healthy from an HIV perspective
  * Patients must have an undetectable HIV viral load
* Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients who have undergone major surgery must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class 2B or better
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of 7+3 treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months). Female patients of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication. Male patients with female partners of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy

  * NOTE: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients with a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Prior treatment with the following are not allowed:

  * Patients who have received anthracyclines for treatment of a prior, unrelated, curatively-treated malignancy which would limit their ability to receive 7 + 3 chemotherapy treatment on study
  * Anti-PD-1, anti-PD-L1, or anti-PD-L2, for a prior, unrelated, curatively-treated malignancy, within last 3 months of enrollment in the study
  * Anti-cancer monoclonal antibody (mAb) within 4 weeks, for a prior, unrelated, curatively-treated malignancy, prior to study registration or have not recovered (recovery defined as baseline or =< grade 1) from AEs due to agents administered more than 4 weeks earlier
  * Experimental treatment within 4 weeks prior to study registration
* Patients who have had chemotherapy (except hydroxyurea and all trans retinoic acid [ATRA] which are allowed but have to be stopped the day before induction therapy starts), targeted small molecule therapy (aside from imatinib, dasatinib, or nilotinib), or curative-intent radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C), for a prior curatively treated malignancy, prior to entering the study
* Patients who have received prior anthracyclines not to exceed 150 mg/m^2 of daunorubicin or equivalent for treatment of a prior, unrelated, curatively-treated malignancy which would limit their ability to receive 7 + 3 chemotherapy treatment on study
* Patients with a cardiac ejection fraction less than 50% as determined by echocardiogram or radionuclide ventriculogram scan (MUGA) scan
* Other active primary malignancy (other than non-melanomatous skin cancer or carcinoma in situ of the cervix) requiring treatment or limiting expected survival to =< 2 years

  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy for their cancer)
* Patients who have FLT3-mutated AML

  * FLT3-ITD or TKD mutations are defined as a mutation with a ratio of mutant to wild-type allele >= 0.05 or variant allele fraction of >= 5% by polymerase chain reaction (PCR) or next generation sequencing from either bone marrow or peripheral blood
  * Note 1: FLT3, karyotype, or FISH results from bone marrow or peripheral blood that were performed up to 3 weeks before initiation of trial therapy are acceptable for eligibility determination or therapy stratification as long as they are performed in a Clinical Laboratory Improvement Act (CLIA) certified laboratory. Note 2: Patients are stratified based on age (younger than 65 versus [vs] 65 and older), presence of core-binding abnormalities by FISH or karyotype (yes/no), and by having t- AML or AML arising from prior/antecedent MDS (yes/no)
* Patients who have not recovered from AEs due to prior anti-cancer therapy (i.e., have not returned to baseline or have residual toxicities > grade 1) with the exception of =< grade 2 neuropathy and alopecia

  * NOTE: Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-CNS disease
* Patients currently participating and receiving study therapy or have participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment are ineligible
* History of hypersensitivity to pembrolizumab (MK-3475) or any of its excipients, or other agents used in this study
* Current use of corticosteroids

  * EXCEPTION: Low doses of steroids (< 10 mg of prednisone or equivalent dose of other steroid) used for treatment of non-hematologic medical condition (e.g., chronic adrenal insufficiency) is permitted
* Patients who underwent prior allogenic transplant
* Patient with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Patient with known active CNS disease and/or carcinomatous meningitis before study enrollment. Assessment of the cerebral spinal fluid (CSF) is not required to enroll in the study unless there is clinical suspicion for CNS involvement. However, if CSF assessment is performed for any reason, there should be no evidence of active leukemia in the CSF as per investigator judgement. Up to one dose of prophylactic intrathecal chemotherapy is allowed prior to study enrollment. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of protocol treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to protocol treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Patients with active autoimmune disease except for patients with hypothyroidism and vitiligo that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients with a known history of non-infectious pneumonitis that required the use of steroids or current pneumonitis
* Patients with active, uncontrolled infection as deemed by the treating investigator
* Patients with a known history of active TB (Bacillus tuberculosis)
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because pembrolizumab (MK-3475) is humanized antibody with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab (MK-3475), breastfeeding should be discontinued if the mother is treated with pembrolizumab (MK-3475). These potential risks may also apply to other agents used in this study
* Patient who have received a live vaccine within 30 days of planned start of study therapy

  * NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist [registered trademark]) are live attenuated vaccines, and are not allowed
* Active hemolytic anemia requiring immunosuppressive therapy or other pharmacologic treatment. Patients who have a positive Coombs test but no evidence of hemolysis are NOT excluded from participation
* Patients with clinically significant disseminated intravascular coagulation (DIC), which cannot be managed with supportive care including transfusions, as assessed by treating physician, will be excluded from study
* Patients with no bone marrow involvement will be excluded (i.e., those with only extramedullary disease)
* Patients with acute promyelocytic leukemia will be excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Rate of minimal residual disease (MRD) negative - complete response (CR)/complete remission with incomplete recovery (CRi) | At time of count recovery after first cycle of consolidation therapy with chemotherapy and pembrolizumab
  MRD will be assessed by multicolor flow cytometry at a central laboratory as an integral biomarker.
Rate of MRD-negative CR | At end of induction therapy
Rate of MRD-negative CR | At end of consolidation

SECONDARY OUTCOMES:
Rate of CR/CRi | At time of count recovery after induction therapy with chemotherapy and pembrolizumab
  Will be defined per European LeukemiaNet 2017.
MRD negativity | At day 14
Rates of complete remission with partial recovery count and hematologic improvement to red blood cells and platelets | Up to end of maintenance
Percentage of patients with MRD-CR using a MRD cutoff of 0.01% | At time of count recovery after first cycle of consolidation therapy
Event-free survival | From randomization to failure to achieve CR/CRi, relapse or death from any cause, assessed up to 5 years
Relapse-free survival (RFS) | From first documentation of CR/CRi to either disease relapse or death from any cause, assessed up to 5 years
  Median RFS will be estimated with Kaplan-Meier curves with 95% confidence interval calculated based on the Brookmeyer-Crowley method
Duration of response (DOR) | From first CR to the date of the first documented relapse or death, whichever occurs first, assessed up to 5 years
  Median DOR will be estimated with Kaplan-Meier curves with 95% confidence interval calculated based on the Brookmeyer-Crowley method.
Incidence of adverse events | Up to 35 days from start of treatment
  Will be assessed per Common Terminology Criteria for Adverse Events version 5.0.

OTHER OUTCOMES:
MRD assessment | Up to end of consolidation
  Will be assessed by duplex sequencing. Library preparation, sequencing, and analysis will be performed with TwinStrand's optimized workflow, and TwinStrand's bioinformatics core will perform all analyses related to assay output.
MRD detection | Up to end of consolidation
  Will compare duplex sequencing and multiparameter flow cytometry for MRD detection. McNemar's Chi-squared test for paired samples (regular duplex sequencing versus multiparameter flow cytometry and ultra-deep duplex sequencing versus multiparameter flow cytometry) will be used to compare the MRD measures.
Immune cell subsets | At time of relapse, assessed up to 3 years
  Will assess immune cell subsets and correlate with response to combine chemotherapy and anti PD-1 directed therapy using mass cytometry. All data will be analyzed and graphs generated using the DVS Cytobank software (Cytobank). Will also measure CD47 levels on leukemic blasts prior to and after chemotherapy and pembrolizumab application to see whether CD47 expression levels correlate with responders versus non-responders and whether expression levels change at different times of therapy. Statistical analyses of the frequency of CD8 positive (+), CD4+, Foxp3 T regulatory cells (Tregs), CD8+/Foxp3+ Tregs, central memory effector (TCM)/ memory cells that re-express CD45RA (TEMRA), effector memory (TEM)/TEMRA, the percentage of Ki67 and GzmB in PD-1+, Eomes+ CD8 T-cells to compare changes over time from baseline to several time-points will be performed by using mixed effects modeling with a Benjamini-Hochberg correction to control for false discovery rates.
PD-1 and PD-L1 expression | At time of relapse, assessed up to 3 years
  An association of clinical response with the expression of PD-L1 acute myeloid leukemia bone marrow cells will be assessed by a Pearson Chi-square test on a 2 x 2 table of frequencies. The dependent variable will be defined as response (yes versus no), and quantitative immunofluorescence categories (negative versus positive) will be the independent variables. Will also monitor the dynamic change of PD-L1 expression over the course of treatment and its correlation with clinical response. Longitudinal measurements of PD-L1 will be examined using mixed-effects modeling.
Genomic deoxyribonucleic acid (DNA) of tumor cells | Baseline
  Will use massively parallel sequencing technology to sequence the genomic DNA of tumor cells (leukemic bone marrow) and normal cells (germline) obtained from patients with acute myeloid leukemia. Mutational load by whole-exome sequencing will be correlated with clinic-pathological parameters such as response to treatment, survival and immune infiltrating profile, and T cell repertoire diversity and clonality.
Protein signatures | At time of relapse, assessed up to 3 years
  Will investigate protein signatures associated with response and efficacy using the Olink inflammation biomarker panel.
Ribonucleic acid (RNA) integrity of formalin fixed paraffin-embedded RNA | Up to time of relapse, assessed up to 3 years
  Will be assessed using either the Agilent 4200 TapeStation and High Sensitivity RNA ScreenTape or the Agilent 2100 Bioanalyzer and RNA 6000 Pico Chip. Either method will employ the region analysis method to determine the percentage of RNA in the sample that is > 200 nt for each sample to be processed.
T cell receptor (TCR) sequencing | Up to time of relapse, assessed up to 3 years
  Will perform high-throughput sequencing of the TCR V beta CDR3 regions on ﬂow cytometrically sorted T-cell subsets to assess the effect of immunotherapy on the diversity of the T-cell repertoire and assess for correlation to clinical outcomes. TCR diversity and clonality will be calculated using a software by Adaptive Technologies. T-cell repertoire diversity and clonality will be correlated with clinic-pathological parameters such as response to treatment, survival, and immune infiltrating profile, as well as genomic profiles (total mutation burden, non-synonymous mutation burden, predicted neoantigen burden, clonal mutation burden and clonal predicted neoantigen burden). TCR profile generated from treatment-refractory tumors at the time of disease progression will be compared to data from pre-treatment tumor samples to explore the TCR repertoire evolution of these tumors under therapeutic pressure.
Gut microbiome | At time of post-consolidation cycle 1
  Analysis of microbiome communities will be performed in R. Pairwise differences in temporal variability across body sites will be made using Mann-Whitney U test, whereas pairwise differences among response groups performed using Student's t-test. Correlation between microbial/metabolome changes with immune-checkpoint expression and kinetics of immune cell subset recovery and programming in the standard of care and experimental arm will be evaluated. As a marker of mucosal immunity, changes in immune cell content within stool samples in patients that experience colitis or gastrointestinal graft versus host disease will be compared to suitable controls.

CONTACTS AND LOCATIONS:
Overall Officials: Amer M Zeidan, Principal Investigator — Yale University Cancer Center LAO
Locations (10):
- United States (10):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04214249/ICF_000.pdf